CLINICAL TRIAL: NCT03169478
Title: The Efficacy of Intrauterine Balloon Dilatation Therapy in the Prevention of Adhesion Formation After Hysteroscopicremovalof Multiple Fibroids
Brief Title: Intrauterine Balloon Dilatation Therapy in the Prevention of Adhesion Formation After Hysteroscopic Myomectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fu Xing Hospital, Capital Medical University (Other)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Xiaoyu Shi, Principal Investigator, Fu Xing Hospital, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017FXHEC-KY005
Record Dates: First submitted 2017-05-25; First posted 2017-05-30 (Actual); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Intrauterine Adhesion
Keywords: hysteroscopic myomectomy; balloon dilatation; adhesions
MeSH Terms: conditions — Gynatresia; Tissue Adhesions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- multiple myoma control group (No Intervention): The control group will not have any balloon therapy. A second-look hysteroscopy will be carried out 6 weeks after the surgery.
- multiple myoma IUB dilatation group (Experimental): The multiple myoma study group will have Foley-catheter intrauterine balloon dilatation therapy 2 weeks and 4 weeks after hysteroscopic myomectomy. A second-look hysteroscopy will be carried out 6 weeks after the surgery.
  Interventions: Procedure: multiple myoma IUB dilatation group

INTERVENTIONS:
Procedure: multiple myoma IUB dilatation group — A Foley catheter (size 8-12fr) will be prepared by cutting the excess catheter tip protruding beyond the balloon. Once the catheter has reached the fundus, 3-5mls of saline will be slowly introduced into the balloon under ultrasound guidance, in order to directly visualize the distention of the cavity and stretching and blunt dissection of any intrauterine adhesions, if present.
  Arms: multiple myoma IUB dilatation group

SUMMARY:
Transcervical resection of submucous myomas (TCRM) is nowadays considered necessary if it is associated with infertility or miscarriage or menorrhagia. Nevertheless, one possible risk of hysteroscopic myomectomy is the formation of intrauterine adhesion (IUA) at the site of resection. The development of IUA arising from trauma to the basalis layer of the endometrium during hysteroscopy can result in infertility, recurrent miscarriages, amenorrhea, dysmenorrhea, or abnormal placentation.

Several measures have been proposed in an effort to decrease the formation of post-surgical intrauterine adhesions. Additionally, physical barriers such as balloon catheters or intrauterine devices have been used in the postoperative period. Despite years of studies evaluating prevention strategies for intrauterine adhesion formation after operative hysteroscopy, it is still unclear which strategy is most effective because there has never been any formal properly powered randomized, control trial to examine the efficacy of the various methods used to prevent adhesion reformation.

In this prospective, randomized, controlled study, the investigators wish to examine the efficacy of intrauterine balloon dilatation therapy in the early postoperative period in preventing adhesion formation after transcervical resection of submucous myomas.

DETAILED DESCRIPTION:
Objectives

To investigate the efficacy of intrauterine balloon (IUB) dilatation therapy in the prevention of adhesion formation after transcervical resection of submucous myomas (TCRM).

Patients

The patients will be recruited from two centers, namely, the Hysterscopy Center of the Fuxing Hospital and TianTan Hospital, Capital Medical University, Beijing, China. Before the surgery all patients with suspected submucous myomas will undergo preoperative evaluations including trans-vaginal ultrasonography. The inclusion criteria include [1] women aged 18-45 years with regular 25-35 days cycles ; [2] no evidence of intrauterine adhesions at the time of surgery; [3] written consent obtained; and [4] agreement to have second-look hysteroscopy; [5] had more than one fibroids removed at the time of hysteroscopic surgery. The exclusion criteria include women who are already postmenopausal or women who have evidence of intrauterine adhesions at the time of surgery.

Study Design

After the completion of transcervical resection of submucous myomas (TCRM), recruited patients will be randomized to one of the two treatment groups by computer-generated numbers: [1] study group will have Foley-catheter intrauterine balloon dilatation therapy 2 weeks and 4 weeks after hysteroscopic myomectomy; [2] the control group will not receiveany balloon therapy. A second-look hysteroscopy will be carried out around 6 weeks after the surgery.

Procedure

Surgical procedure

The surgery will be carried out by an experienced hysteroscopic surgeons with the use of a 8.5 mm rigid hysteroscope with under 100-120 mm Hg pressure. The procedure will be performed under general anesthesia in a day surgery unit under ultrasonographic guidance. Once the type and number of myomas have been verified, the myoma will be then be bluntly dissected from the muscular layer with the tip of the resectoscope. After the myomas have been dissected from the muscular layer, they will be shaved into pieces to reduce the volume and then be retrieved from the uterine cavity with a myoma grasper.

Postoperative treatments

All patients will be treated with oral antibiotics for 3-5 days in line with local practice. Second-look hysteroscopy will be carried out 6 weeks after the initial operation. After assessment of the extent and severity of any newly formed adhesion, hysteroscopic adhesiolysis, if needed, will be carried out at the time of the second-look procedure. Immediately prior to second look hysteroscopy, a swab will be taken from the endo-cervical canal for routine bacteriological study; At the conclusion of the second look hysteroscopy, an endometrial sample will be obtained for histological study &immune histochemical analysis including evidence of chronic endometrtitis(CD138 staining). The surgeons who perform the second-look will be blinded to the randomization.

IUB dilatation therapy

IUB dilatation therapy will be performed according to the methodology published in the literature. In brief, a Foley catheter (size 12-14fr) will be prepared by cutting the excess catheter tip protruding beyond the balloon. Once the catheter has reached the fundus, 3-5mls of saline will be slowly introduced into the balloon under ultrasound guidance, in order to directly visualize the distention of the cavity and stretching and blunt dissection of any intrauterine adhesions, if present.

Statistical Analysis

The efficacy of treating the intrauterine adhesions in the two groups will be compared using the χ2 test. The AFS score in the two groups will be compared using the Mann-Whitney U test. A p value of < 0.05 will be considered statistically significant. All statistical analysis will be carried out with the use of SPSS 21.0.

Power calculation

On the basis of the investigators own internal audit and the results of the two published retrospective cohort studies analysing the prevalence of intrauterine adhesion (IUA) formation in women undergoing transcervical resection of multiple submucousmyomas (TCRM),the investigators estimated that the adhesion formation rate in the control group to be 25% and the treatment group (balloon group) to be 5%; accepting a type 1 error of 0.05, and a type 2 error of 0.10, the number of subjects required in each arm of the randomized controlled trial would be 51. Assuming that the drop-out rate to be 10%, the total number of subject to be recruited would be 56 in each arm, that is a total of 112.

Outcome measures

The primary outcome measure will be the amount of intrauterine adhesions as measured according to the AFS score at follow-up. The secondary outcome measures will include any complications including any clinical infection and change of menstrual pattern after surgery and the need for re-operation.

Data processing and analysis

The researchers will ensure the confidentiality of sensitive data by minimizing the number of personnel who handle subject data. In addition, computer data will be encrypted as required to maximize security, while paper documents will be locked in filing cabinets, with only authorized personnel having access to the information.

Ethical considerations

IUB dilatation has been published as a novel technique with no untoward complications identified to date. The procedure will be performed according to the methodology available in the literature and the study has gained approval from the local ethical committee (Approval Notice Number:2016FXHEC-KY005).

Consent

All subjects will be given a detailed explanation of the study and sufficient time to consider participants. A written consent form will be signed by the patient and retained in the investigators confidential records.

ELIGIBILITY:
Inclusion Criteria:

* [1] women aged 18-45 years with regular 25-35 days cycles ;
* [2] no evidence of intrauterine adhesions at the time of surgery;
* [3] written consent obtained;
* [4] agreement to have second-look hysteroscopy;
* [5] had more than one fibroids removed at the time of hysteroscopic surgery

Exclusion Criteria:

* [1] women who are already postmenopausal
* [2] women who have evidence of intrauterine adhesions at the time of surgeryare

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The study focus on intrauterine adhesion only in female patients.
Enrollment: 112 (Estimated)
Dates: Start 2017-05-30 (Actual); Primary Completion 2019-05-30 (Estimated); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
The amount of intrauterine adhesions at second look hysteroscopy | at 6 weeks post-op
  The amount of intrauterine adhesions according to AFS score at second look hysteroscopy

SECONDARY OUTCOMES:
complications of hysteroscopic myomectomy | at 6 weeks post-op
  complications of hysteroscopic myomectomy including infection rate
menstrual pattern | at 3 months post-op
  The menstrual pattern before and after surgery and the need for re-operation

CONTACTS AND LOCATIONS:
Overall Officials: Tinchiu Li, Study Chair — Fu Xing Hospital, Capital Medical University
Locations (1):
- Fu Xing Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Saravelos SH, Li TC. Ultrasound-guided treatment of intrauterine adhesions in the outpatient setting. Ultrasound Obstet Gynecol. 2017 Aug;50(2):278-280. doi: 10.1002/uog.16218. No abstract available. PMID 27420903
- [Result] Saravelos SH and Li TC. Intrauterine balloon therapy: a novel ultrasound guided treatment for intrauterine adhesions. Gynecological Surgery [Epub ahead of print]
- [Result] Saravelos SH, Jayaprakasan K, Ojha K, Li TC. Assessment of the uterus with three-dimensional ultrasound in women undergoing ART. Hum Reprod Update. 2017 Mar 1;23(2):188-210. doi: 10.1093/humupd/dmw040. PMID 28007752
- [Result] March CM. Intrauterine adhesions. Obstet Gynecol Clin North Am. 1995 Sep;22(3):491-505. PMID 8524533
- [Result] Orhue AA, Aziken ME, Igbefoh JO. A comparison of two adjunctive treatments for intrauterine adhesions following lysis. Int J Gynaecol Obstet. 2003 Jul;82(1):49-56. doi: 10.1016/s0020-7292(03)00030-4. PMID 12834941
- [Result] Varasteh NN, Neuwirth RS, Levin B, Keltz MD. Pregnancy rates after hysteroscopic polypectomy and myomectomy in infertile women. Obstet Gynecol. 1999 Aug;94(2):168-71. doi: 10.1016/s0029-7844(99)00278-1. PMID 10432121
- [Result] Taskin O, Sadik S, Onoglu A, Gokdeniz R, Erturan E, Burak F, Wheeler JM. Role of endometrial suppression on the frequency of intrauterine adhesions after resectoscopic surgery. J Am Assoc Gynecol Laparosc. 2000 Aug;7(3):351-4. doi: 10.1016/s1074-3804(05)60478-1. PMID 10924629
- [Result] Yang JH, Chen MJ, Wu MY, Chao KH, Ho HN, Yang YS. Office hysteroscopic early lysis of intrauterine adhesion after transcervical resection of multiple apposing submucous myomas. Fertil Steril. 2008 May;89(5):1254-1259. doi: 10.1016/j.fertnstert.2007.05.027. Epub 2007 Aug 8. PMID 17686478
- [Result] Touboul C, Fernandez H, Deffieux X, Berry R, Frydman R, Gervaise A. Uterine synechiae after bipolar hysteroscopic resection of submucosal myomas in patients with infertility. Fertil Steril. 2009 Nov;92(5):1690-3. doi: 10.1016/j.fertnstert.2008.08.108. Epub 2008 Oct 19. PMID 18937941
- [Result] Healy MW, Schexnayder B, Connell MT, Terry N, DeCherney AH, Csokmay JM, Yauger BJ, Hill MJ. Intrauterine adhesion prevention after hysteroscopy: a systematic review and meta-analysis. Am J Obstet Gynecol. 2016 Sep;215(3):267-275.e7. doi: 10.1016/j.ajog.2016.05.001. Epub 2016 May 10. PMID 27173082
- [Result] Guida M, Acunzo G, Di Spiezio Sardo A, Bifulco G, Piccoli R, Pellicano M, Cerrota G, Cirillo D, Nappi C. Effectiveness of auto-crosslinked hyaluronic acid gel in the prevention of intrauterine adhesions after hysteroscopic surgery: a prospective, randomized, controlled study. Hum Reprod. 2004 Jun;19(6):1461-4. doi: 10.1093/humrep/deh238. Epub 2004 Apr 22. PMID 15105384
- [Result] Roge P, D'Ercole C, Cravello L, Boubli L, Blanc B. Hysteroscopic management of uterine synechiae: a series of 102 observations. Eur J Obstet Gynecol Reprod Biol. 1996 Apr;65(2):189-93. doi: 10.1016/0301-2115(95)02342-9. PMID 8730623
- [Result] Schenker JG. Etiology of and therapeutic approach to synechia uteri. Eur J Obstet Gynecol Reprod Biol. 1996 Mar;65(1):109-13. doi: 10.1016/0028-2243(95)02315-j. PMID 8706941
- [Result] Pabuccu R, Atay V, Orhon E, Urman B, Ergun A. Hysteroscopic treatment of intrauterine adhesions is safe and effective in the restoration of normal menstruation and fertility. Fertil Steril. 1997 Dec;68(6):1141-3. doi: 10.1016/s0015-0282(97)00375-0. PMID 9418714